CLINICAL TRIAL: NCT06449313
Title: A Phase 2 Single-Arm Study of Neoadjuvant Chemo-Immunotherapy and Surgical Resection in Locally Advance Non-Small Cell Lung Cancer (NSCLC) With N3 Lymph Node Involvement
Brief Title: Neoadjuvant Chemo-Immunotherapy and Surgical Resection in Locally Advanced Non-small Cell Lung Cancer With N3 Lymph Node Involvement
Acronym: NEO-SURG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007668
Record Dates: First submitted 2024-06-03; First posted 2024-06-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer Stage III
Keywords: non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cemiplimab plus chemotherapy (Experimental): cemiplimab given with standard of care chemotherapy for 4 treatments/cycles before surgery and then every 3 weeks for 1 year after surgery.
  Interventions: Drug: Cemiplimab-Rwlc

INTERVENTIONS:
Drug: Cemiplimab-Rwlc — 350 mg every 3 weeks, intravenously, on day 1 of a 21 day cycle for 4 cycles, then every 3 weeks after surgery for 1 year.
  Other Names: Libtayo

SUMMARY:
The goal of this clinical trial is to learn about neoadjuvant cemiplimab with histology-specific chemotherapy followed by resection and adjuvant cemiplimab in stage 3 non-small cell lung cancer (NSCLC) with contralateral mediastinal or ipsilateral supraclavicular lymph node (N3) involvement..

The main question it aims to answer is whether patients with stage 3 NSCLC with involvement of lymph nodes can undergo surgery to remove the cancer after receiving treatment with chemotherapy + immunotherapy.

Participants will receive FDA-approved chemotherapy called platinum-doublet chemotherapy together with an immunotherapy drug targeting the immune marker PD-1 called cemiplimab. Patients will receive a 3 drug combination for 4 total treatments given every 3 weeks before surgery. After surgery, patients will have the option to undergo radiation therapy if it is recommended by their treatment team. After this, they will receive cemiplimab every 3 weeks for one year.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at time of signing the informed consent form (ICF).
2. Histologically or cytologically confirmed stage 3 B/C Non-Small Cell Lung Cancer (NSCLC) as assessed per the 8th American Joint Committee on Cancer (AJCC) with pathologically-confirmed contralateral mediastinal or ipsilateral supraclavicular (N3) lymph node involvement.
3. Primary tumor appropriate for resection with curative intent as assessed by the treating surgeon prior to study enrollment.
4. Absence of major associated pathologies and co-morbidities that elevate surgery risk to a prohibitive level, as assessed by treating surgeon prior to study enrollment.
5. Pulmonary function capacity capable of tolerating the lung resection proposed by the treating surgeon.
6. EGFR, ALK, wild-type assessed via any CLIA-certified tissue testing platform. Documentation of EGFR and ALK status is not required for pure squamous NSCLC histology.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
8. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 21 days prior to initiation of study treatment:

   1. Absolute Neutrophil count (ANC) ≥ 1.0 x 10^9/L (1000/uL) without granulocyte colony-stimulating factor support
   2. Platelet count ≥ 100 x 10^9/L (100,000/uL) without transfusion
   3. Hemoglobin ≥ 90 g/L (9.0 g/dL) (Patients may be transfused to meet this criterion.)
   4. Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) </= 3 x upper limit of normal (ULN)
   5. Serum bilirubin </= 2.0 x ULN with the following exception: Patients with known Gilbert disease: serum bilirubin </= 3 x ULN
   6. Creatinine clearance ≥ 45 mL/min (calculated using the Cockcroft-Gault formula). If creatinine clearance determined by Cockcroft-Gault is <45 mL/min, another appropriate validated formula or 24hr urine collection may be used in consultation with the study PI.
   7. For patients not receiving therapeutic anticoagulation: INR (international normalised ratio) and aPTT (activated partial thromboplastin time) </= 1.5 x ULN. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen defined as clinical stability on unchanged dose of therapeutic anticoagulation for ≥14 days.
9. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs, as defined below:

   Women must remain abstinent or use highly effective contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 4 months after the final dose of study treatment. Women must refrain from donating eggs during this same period.

   A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.

   Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

   The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.
10. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

With a female partner of childbearing potential who is not pregnant, or a female partner who is pregnant, men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for 4 months after the final dose of study treatment. Men must refrain from donating sperm during this this same period.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.

Exclusion Criteria:

1. NSCLC with histology containing any of the following: large cell neuroendocrine carcinoma, small cell lung cancer.
2. Primary tumor not deemed appropriate for surgical resection as assessed by treating surgeon.

   1. Tumor with direct invasion of: mediastinum, diaphragm, heart, great vessels, trachea, esophagus, vertebral body, or carina.
   2. Any other tumor characteristic making it not suitable for resection as determined by treating surgeon.
3. Any prior systemic therapy for index lung cancer, including immunotherapy, chemotherapy.
4. History of malignancy requiring systemic therapy within 2 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death as assessed and confirmed by the study PI. (Patients with a history of stage I NSCLC treated with resection or radiotherapy are eligible for inclusion.)
5. Active or history of clinically significant autoimmune disease that, in the opinion of the investigator, could compromise the health and safety of the patient if treated with anti-PD1 immunotherapy. Notable exceptions include:

   1. Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone.
   2. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen.
   3. Active or history of adrenal insufficiency on stable steroid regimen.
   4. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only are eligible for the study provided all of following conditions are met: Disease is well controlled at baseline and requires only low-potency topical corticosteroids; No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency oral corticosteroids within the previous 12 months
6. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
7. Known active tuberculosis.
8. Known history of poorly controlled HIV. Patients living with HIV are allowed to enroll if: (1) they are clinically stable on appropriate highly active anti-retroviral therapy (HAART) with undetectable HIV viral load and CD4 count >350 and (2) the HAART regimen poses no unacceptable interactions with the prescribed anti-cancer therapies.
9. Known history of poorly controlled hepatitis B or hepatitis C

   1. Patients with known hepatitis B (HepBsAg+) who have controlled infection (serum hepatitis B virus (HBV) DNA PCR that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA per local standards and must remain on anti-viral therapy for at least 6 months beyond the last dose of investigational study drug.
   2. Patients who are known hepatitis C virus (HCV) antibody positive (HCV Ab+) who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
10. Severe infection within 3 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection (including COVID-19), bacteremia, or severe pneumonia that, in the opinion of the investigator, may impact patient safety.
11. Prior allogeneic stem cell or solid organ transplantation.
12. Any treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during study treatment or within 5 months after the final dose of study treatment.
13. Significant vascular and cardiovascular disease (e.g., New York Heart Association Class II or greater heart failure, unstable arrhythmia, aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis - including but not limited to myocardial infarction, transient ischemic attack, stroke or unstable angina) within 6 months prior to study treatment initiation.
14. Treatment with systemic immunosuppressive medication (including, but not limited to: corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

    1. Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after PI confirmation has been obtained.
    2. Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
15. Any prior use of an immune checkpoint blockade therapy including agents directed against CTLA-4, PD-1, and PD-L1.
16. History of severe allergic reaction or hypersensitivity to study drug components.
17. Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 6 months after the final dose of study treatment. Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rate | 12 weeks
  Pathologic complete response (pCR): 0% viable tumor in primary tumor and resected lymph nodes.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 1 year
  Defined as imaging response according to RECIST v1.1 (Eisenhauer et al. 2009).
Rate of R0 Resection | 12 weeks
  Rate of R0 Resection: Defined as percentage of patients undergo complete tumor resection with negative margins.
Major pathologic response (MPR) rate | 12 weeks
  MPR Rate: Defined as the percentage of patients with resection specimen that shows ≤10% viable tumor in resected lung and lymph nodes
Disease-free Survival (DFS) | 5 years
  DFS: Time from first dose of neoadjuvant treatment to documented disease recurrence. Where possible, date of pathologic confirmation of recurrence should be used over date of radiographic imaging showing findings concerning for recurrence.
Overall Survival (OS) | 5 years
  Time first dose of neoadjuvant treatment to death.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Reuss, MD, Principal Investigator — Georgetown University
Locations (3):
- United States (3):
  - Lombardi Comprehensive Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - Washington University School of Medicine-Sitemen Cancer Center, St Louis, Missouri
  - UVA Comprehensive Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No